CLINICAL TRIAL: NCT05175430
Title: Effects of Serotonin Transporter Inhibition on the Subjective Response to LSD in Healthy Subjects
Brief Title: Effects of SERT Inhibition on the Subjective Response to LSD in Healthy Subjects
Acronym: SERT-LSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2021-02223
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: LSD; psychedelics; SSRI; healthy subjects; serotonin; 5-HT2A
MeSH Terms: interventions — Paroxetine; Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: 2-period cross-over, randomized, double-blind (paroxetine vs. placebo) study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pretreatment with paroxetine (Active Comparator): Pretreatment with paroxetine (10 mg daily for 1 week followed by 20 mg daily for 5 weeks, per os), followed by administration of LSD (0.1 mg, per os) on the study day
  Interventions: Drug: Paroxetine; Drug: Lysergic Acid Diethylamide
- Pretreatment with placebo (Placebo Comparator): Pretreatment with placebo for 6 weeks (mannitol, per os), followed by administration of LSD (0.1 mg, per os) on the study day
  Interventions: Drug: Lysergic Acid Diethylamide; Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine — Paroxetine (per os) will be used as pharmacological tool to downregulate 5-HT1/2 receptors.
  Arms: Pretreatment with paroxetine
Drug: Lysergic Acid Diethylamide — LSD (per os) will be used to see if 5-HT 1/2 receptors were downregulated by paroxetine.
  Other Names: LSD
Drug: Placebo — Placebo (per os) for the Paroxetine condition will be used to compare the data from the study day with LSD between both arms.
  Arms: Pretreatment with placebo

SUMMARY:
Lysergic acid diethylamide (LSD) is a classic serotonergic psychedelic acting on the serotonin 5-HT2A receptor. LSD is used recreationally and in psychiatric research. First studies suggest efficacy in psychiatric disorders, such as depression and anxiety. SSRIs like paroxetine are first-line treatments for depression and anxiety disorders. Paroxetine acts as a serotonin transporter (SERT) inhibitor. However, the link between this mechanism and its positive effects on mood remains to be established. Several studies suggest a possible downregulation of postsynaptic serotonin (5-HT) receptors such as the 5-HT2A receptor. The aim of the study is to assess whether SERT inhibition reduces expression of the gene coding for the 5-HT2A receptor and the response to LSD.

DETAILED DESCRIPTION:
Participants will be treated with paroxetine (Paroxetine 10 mg daily for 1 week followed by 20 mg daily for 5 weeks) or placebo for 6 weeks. Pretreatment is followed the first study day. A single dose of LSD (0.1 mg) will be administered. Primary study endpoint are the subjective effects on consciousness (5D-ASC total score). Secondary study endpoints include additional psychological measurements, plasma concentrations of LSD and paroxetine, as well as some safety measures (autonomic effects, ECG). The washout between the first study day and the second pretreatment will be at least 2 days. In the second pretreatment period, participants will be treated with placebo or paroxetine (cross-over) for another 6 weeks. This is followed by the second study day and administration of LSD (0.1 mg).

Based on a power analysis the sample size is 24 participants (12 female and 12 male).

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the German language.
* Understanding the procedures and the risks that are associated with the study.
* Participants must be willing to adhere to the protocol and sign the consent form.
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to abstain from xanthine-based liquids from the evenings prior to the study sessions and during the sessions.
* Participants must be willing not to drive a traffic vehicle or to operate machines within 48h after substance administration.
* Willing to use double-barrier birth control throughout study participation.
* Body mass index between 18-29 kg/m2.

Exclusion Criteria:

* Chronic or acute medical condition, including a history of seizures.
* Current or previous major psychiatric disorder (e.g. psychotic disorders, mania / hypomania, anxiety disorders).
* Psychotic disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain.
* Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg); QT-time>450 ms (men) or >470 ms (women).
* Use of hallucinogenic substances (not including cannabis) more than 20 times or any time within the previous two months.
* History of acute glaucoma.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days).
* Use of medications that may interfere with the effects of the study medications (any psychiatric medications and any medication with known pharmacokinetic or pharmacodynamic interactions with paroxetine).
* Tobacco smoking (>10 cigarettes/day).
* Consumption of alcoholic drinks (>20 drinks/week).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
5 dimensions of altered state of consciousness (5D-ASC) total OAV score | Study sessions per participant will be separated by at least 43 days
  Visual analog scale consisting of 94 items. Constructed of five scales and allows assessing mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. Scales will be presented as 100 mm long horizontal lines marked with vertical lines by the participant.
Visual Analog Scales (VAS) good effect rating | Study sessions per participant will be separated by at least 43 days
  VAS will be presented as 100 mm long horizontal lines marked with "not at all" on the left and "extremely" on the right. The following VAS items will be used: "any drug effect", "good drug effect", "bad drug effect", "drug high", "anxiety", "nausea", "feeling depressed", "alteration of vision", "alterations of hearing", "sounds seem to influence what I see", "alteration of sense of time", "the boundaries between myself and my surroundings seem to blur", "I gain insights into contexts that were previously were inscrutable to me", "talkative", "open", "trust" and "the context of my thought is personal/impersonal". Subjects will mark the scale with vertical lines.

SECONDARY OUTCOMES:
Adjective mood rating scale (AMRS) | Study sessions per participant will be separated by at least 43 days
  The adjective mood rating scale (AMRS or EWL60S) is a 60-item Likert scale that allows repeated assessment of mood in 6 dimensions: activation, inactivation, well-being, anxiety/depressed mood, extroversion and introversion, and emotional excitability.The AMRS consists of subscales measuring "activation", "positive mood", "extroversion", "introversion", "inactivation", and "emotional excitability.
States of consciousness questionnaire (SCQ) | Study sessions per participant will be separated by at least 43 days
  This 100-item questionnaire is rated on a six-point scale. Forty-three items embedded into this questionnaire comprise the Mystical Experience Questionnaire (MEQ). which is sensitive to the effects of psilocybin. The 43 items provide scale scores for each of seven domains of mystical experiences: internal unity (pure awareness, a merging with ultimate reality), external unity (unity of all things, all things are alive, all is one), sense of sacredness (reverence, sacred), noetic quality (encounter with ultimate reality, more real than everyday reality), transcendence of time and space, deeply felt positive mood (joy, peace, love), paradoxicality/ineffability (claim of difficulty in describing the experience in words). We will also derived the four scale scores of the newly validated revised 30-item MEQ: mystical, positive mood, transcendence of time and space, and ineffability.
Spiritual Realm Questionnaire (SRQ) | Study sessions per participant will be separated by at least 43 days
  This questionnaire has recently been developed by linguist and psychologist K. Stocker, Swiss Federal Institute of Technology Zürich and University of Zürich, to rate psychedelic (entheogenic) experiences with a focus on spiritual aspects insufficiently covered by the 5D-ASC and SCQ. The scale includes 11 main questions to be answered on a total of 65 sub-ordered visual rating scales. Results will be used to validate the scale and will be analyzed similar to the 5D-ASC using paired t-tests and comparing the constructs defined by the 11 main questions contained within the four main dimensions religious-psychological spirituality spectrum of humanity, human condition and life meaningfulness, dealing with personal problems, and worldview/belief.
Psychological Insight Questionnaire (PIQ) | Study sessions per participant will be separated by at least 43 days
  This is a newly developed instrument to assess the degree to which an event has facilitated acute insight and gained awareness into emotions, behaviors, beliefs, memories, or relationships. The 14 items resulting from a recent validation process are to be rated on a 6-point Likert scale ranging from 0 = "No; not at all" to 5 = "Extremely (more than ever before in my life)".
Blood pressure | Study sessions per participant will be separated by at least 43 days
  Repeatedly measured using blood pressure / pulse apparatus (mmHg scale)
Heart rate | Study sessions per participant will be separated by at least 43 days
  Repeatedly measured using blood pressure / pulse apparatus (beats per minute scale)
Body temperature | Study sessions per participant will be separated by at least 43 days
  Repeatedly measured using ear thermometer (degree Celsius scale)
Plasma concentrations of paroxetine | Study sessions per participant will be separated by at least 43 days
  Paroxetine plasma concentrations will be measured repeatedly over time using LC-MS/MS techniques (nanogram per milliliter scale)
Plasma concentrations of LSD | Study sessions per participant will be separated by at least 43 days
  LSD plasma concentrations will be measured repeatedly over time using LC-MS/MS techniques (nanogram per milliliter scale)
HTR gene expression | Study sessions per participant will be separated by at least 43 days
  Messenger ribonucleic acid (mRNA) expression levels in whole blood as a peripheral marker of spiny neuronal gene (CNS) expression will be used to measure expression of HTR genes as well as expression of the SERT gene.
Changes in the electrocardiogram (ECG) | Study sessions per participant will be separated by at least 43 days
  Corrected QT time (QTc) will be measured twice on the study days (baseline and at peak drug effect) to examine possible drug-induced changes in the ECG as well as a safety measure (millisecond scale).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Dr., MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No